CLINICAL TRIAL: NCT00069810
Title: Oxidative Stress in Chronic Kidney Disease
Brief Title: Role of Chronic Kidney Disease in Cardiovascular Disease
Status: Withdrawn | Type: Observational
Why Stopped: The study is not a clinical trial.
Sponsor: University of Washington (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Jonathan Himmelfarb, MD, Harborview Medical Center
Other Study IDs: 1234; R01HL070938 (NIH)
Record Dates: First submitted 2003-10-01; First posted 2003-10-06 (Estimated); Last update posted 2017-04-06 (Actual); Status verified 2017-04

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Kidney Failure, Chronic
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — EDTA tube of whole blood
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine how the progressive loss of kidney function influences cardiovascular disease.

DETAILED DESCRIPTION:
BACKGROUND:

Currently, both the incidence and prevalence of chronic kidney disease leading to end-stage renal disease (ESRD) continue to increase at an alarming rate in the United States. According to the United States Renal Data System, in 2000 there were 370,000 prevalent ESRD patients, which was expected to grow to 610,000 by the year 2010. Furthermore, the adjusted death rate for all incident ESRD patients was 19.8 per 100 patient years at risk, with cardiovascular disease accounting for more than 50 percent of mortality in this patient population. Recent analyses demonstrate that there are at least 10.9 million people in the United States with chronic kidney disease and, that for this population, there are substantially increased cardiovascular risks, prompting the Surgeon General to include chronic kidney disease as a focus area for improving the nation's health in Healthy People 2010. The metabolic derangements accompanying progressive loss of kidney function lead to unique patterns of oxidative injury specific to the uremic state. For patients with chronic kidney disease, non-traditional risk factors for cardiovascular disease such as increased oxidative stress and inflammation may be especially important.

DESIGN NARRATIVE:

The broad goals of this study are to develop enhanced understanding of how the progressive loss of kidney function leads to increased oxidative stress, inflammation, and accelerated development of cardiovascular disease. The long-term objective of this proposal is to develop the data critical for a subsequent large scale, multicenter, randomized, controlled trial designed to alleviate oxidative stress, reduce inflammation, and reduce cardiovascular morbidity in patients with chronic kidney disease. The aims of this study are to determine in a prospective study the extent to which oxidative stress is a risk factor for cardiovascular events in patients with chronic kidney disease and to characterize the inter-relationships between oxidative stress and inflammation. A further aim is to determine in the longitudinal study is how progressive loss of kidney function influences oxidative stress propensity to inflammation and cardiovascular disease. An additional aim is to determine the effects of antioxidant therapy on biomarkers of oxidative stress, markers of inflammation and endothelium-dependent vascular function in patients with chronic kidney disease. This study incorporates a series of observational and interventional studies measuring the extent of cardiovascular disease with extensive ex vivo measures of biomarkers of oxidative stress and inflammation in patients with chronic kidney disease. Coordination between the clinical data and the ex vivo studies will be emphasized to achieve maximal understanding of the pathophysiology of uremic cardiovascular disease.

ELIGIBILITY:
Inclusion Criteria:

* Mentally competent and willing to sign the consent form
* Agree to follow up with our nephrology clinic every 3 months for 3 years
* Agree to have the carotid Doppler studies, transthoracic echocardiogram, and brachial artery Doppler measurements

Exclusion Criteria:

* Do not wish to participate
* Acute inflammatory illness
* On experimental drug protocols
* Hypersensitivity to organic nitrates, isosorbide, or nitroglycerin
* Pregnant women
* Atrial fibrillation (only for those undergoing pulse wave velocity)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: People with chronic kidney disease and healthy subjects
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2003-08; Primary Completion 2010-12 (Estimated); Study Completion 2010-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Himmelfarb, MD, Principal Investigator — Harborview Injury Prevention and Research Center

REFERENCES:
- [Background] Simmons EM, Langone A, Sezer MT, Vella JP, Recupero P, Morrow JD, Ikizler TA, Himmelfarb J. Effect of renal transplantation on biomarkers of inflammation and oxidative stress in end-stage renal disease patients. Transplantation. 2005 Apr 27;79(8):914-9. doi: 10.1097/01.tp.0000157773.96534.29. PMID 15849543